CLINICAL TRIAL: NCT03429179
Title: Using Pre-operative Anxiety Score to Determine the Precise Dose of Butorphanol in Patients Undergoing Orthopedic Procedures: A Double-blinded Randomized Trial
Brief Title: Using Preoperative Anxiety Score to Determine the Precise Dose of Butorphanol for Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: the effect of butorphanol
Record Dates: First submitted 2018-01-20; First posted 2018-02-12 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-03

CONDITIONS: Preoperative Anxiety; Precise Dose of Butorphanol
Keywords: butorphanol; preoperative anxiety; sedation; recommend dose
MeSH Terms: interventions — Butorphanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High anxiety butorphanol group (Experimental): preoperative anxiety score of Amsterdam pre-operative anxiety and information scale(APAIS) in high anxiety butorphanol group were >10，and received an intravenous loading dose of 15ug/kg butorphanol 5 mins before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion when the Ramsay sedation score (RSS) reached 4
  Interventions: Drug: Butorphanol
- High anxiety 0.9% saline group (Placebo Comparator): preoperative anxiety score of Amsterdam pre-operative anxiety and information scale(APAIS) in high anxiety 0.9% saline group were >10, and received an infusion of the same volume of 0.9% saline
  Interventions: Other: Physiological saline
- Low anxiety butorphanol group (Experimental): preoperative anxiety score of Amsterdam pre-operative anxiety and information scale(APAIS) in low anxiety butorphanol group were ≤10,and received an intravenous loading dose of 15ug/kg butorphanol 5 mins before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion when the Ramsay sedation score (RSS) reached 4
  Interventions: Drug: Butorphanol
- Low anxiety 0.9% saline group (Placebo Comparator): preoperative anxiety score of Amsterdam pre-operative anxiety and information scale(APAIS) in low anxiety 0.9% saline group were ≤10, and received an infusion of the same volume of 0.9% saline
  Interventions: Other: Physiological saline

INTERVENTIONS:
Drug: Butorphanol — intravenous loading dose of 15ug/kg butorphanol 5 mins before starting the surgery, then followed by infusion of 7.5ug/kg/h butorphanol and stopped infusion when the Ramsay sedation score (RSS) reached 4
  Arms: High anxiety butorphanol group; Low anxiety butorphanol group
Other: Physiological saline — intravenous infusion of the same volume of 0.9% saline
  Arms: High anxiety 0.9% saline group; Low anxiety 0.9% saline group

SUMMARY:
Pre-operative anxiety usually lead to increased anesthetics during the surgery. The precise sedative requirement which can keep adequate sedative state and avoid adverse effects caused by excessive drugs still needs further study. Therefore, our purpose was to confirm the sedative effect of butorphanol and to explore the relationship between pre-operative anxiety and intra-operative butorphanol requirement to evaluate the precise sedative requirement which can keep adequate sedation for patients by pre-operative anxiety score.

DETAILED DESCRIPTION:
A total of 142 patients (aged 18-75 years) who were scheduled for elective low limb orthopedic procedures under spinal anesthesia were included in this study. Patients were divided into two groups based on pre-operative anxiety score evaluated by the Amsterdam pre-operative anxiety and information scale before the surgery. And intramuscular midazolam 0.05mg/kg as a premedication in preoperative room was given to patients before shifting into operation room. Patients in each group were randomly divided into butorphanol group and 0.9% saline group. The sedation score, the duration of reaching adequate sedation state and postoperative recovery were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ-Ⅱ
* age 18-75 years
* surgical operation of lower extremities in orthopedics
* no contraindication of epidural anesthesia

Exclusion Criteria:

* with central system disease
* with cardiovascular disease
* with autonomic nervous system disease
* long term use of analgesic drugs ,sedative drugs,and anti-anxiety drugs
* language barrier
* unwilling to cooperate with the experimenter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety score assessed by the Amsterdam preoperative anxiety and information scale (APAIS)". | before the surgery
  evaluate the preoperative anxiety score before the surgery, APAIS contains 6 items rated on a five-point Likert scale, which represents two scales: anxiety (items 1, 2, 4, and 5) and need for information (items 3 and 6) Accordingly, the maximal score of the entire APAIS (APAIS-T) is 30 and the one expressing the patient's need for information (APAIS-I) is 10. The maximal score of the two items concerning anxiety about anesthesia (APAIS-A-An) and surgery (APAIS-A-Su) is also 10 each, resulting in a maximal score of 20 for total preoperative anxiety (APAIS-A-T). And APAIS-A-T > 10 was used as a cut-oﬀ to deﬁne patients with high anxiety, the higher the score, the more serious the pre-operative anxiety is
Ramsay Sedation score | during the surgery
  evaluate the Ramsay sedation score 10min after getting into the operation room and 5,10,15,30min after infusion.The Ramsay Sedation score ranges from 1-6. 1, anxious and agitated or restless or both; 2, cooperative, orientated, and tranquil; 3, responds to commands only; 4, brisk response to a light glabellar tap or auditory stimulus; 5, sluggish response to a light glabellar tap or auditory stimulus; and 6, no response to a light glabellar tap or auditory stimulus
The time when Ramsay sedation score reached 4 points | Ramsay sedation score reach 4 points during the surgery
  record the time when Ramsay sedation score reached 4 points.The Ramsay Sedation score ranges from 1-6. 1, anxious and agitated or restless or both; 2, cooperative, orientated, and tranquil; 3, responds to commands only; 4, brisk response to a light glabellar tap or auditory stimulus; 5, sluggish response to a light glabellar tap or auditory stimulus; and 6, no response to a light glabellar tap or auditory stimulus
vital signs | during the surgery
  Record Mean Arterial Pressure(MAP)10min after getting into the operation room and 5,10,15,30min after infusion

SECONDARY OUTCOMES:
vital signs | during the surgery
  Record SPO2 10min after getting into the operation room and 5,10,15,30min after infusion
Vital signs | during the surgery
  Record Heart Rate(HR) 10min after getting into the operation room and 5,10,15,30min after infusion
The incidence of nausea/vomiting dizzy bradycardia and hypotension | first day after the surgery
  investigate the incidence of nausea/vomiting dizzy bradycardia and hypotension in the first day after the surgery
post operative visual analgesia scale scores (VAS) | within 24 hours after the surgery
  assess the visual analgesia scale scores (VAS) every hour till 6 h and then every 2 h till 24 h
postoperative patient satisfaction | first day after the surgery
  Patient satisfaction was recorded on 5 levels: a) agreeable experience; b) neither pleasant nor unpleasant; c) slightly uncomfortable; d) disagreeable; e) a traumatic experience.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu junchao, doctor, Study Director — Shengjing Hospital
Locations (1):
- shengjing hospital of China medical university, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Song B, Yang Y, Teng X, Li Y, Bai W, Zhu J. Use of pre-operative anxiety score to determine the precise dose of butorphanol for intra-operative sedation under regional anesthesia: A double-blinded randomized trial. Exp Ther Med. 2019 Nov;18(5):3885-3892. doi: 10.3892/etm.2019.8040. Epub 2019 Sep 23. PMID 31611935